CLINICAL TRIAL: NCT00507494
Title: Influence of Pioglitazone for Renal Transplant Function in Diabetics - a Double Blind Randomised Placebo Controlled Cross Over Study
Brief Title: Influence of Pioglitazone for Renal Transplant Function in Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DNTx
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Diabetes Mellitus; Kidney Transplantation; Proteinuria
Keywords: posttransplant diabetes mellitus; kidney transplantation; filtration fraction; proteinuria
MeSH Terms: conditions — Diabetes Mellitus; Proteinuria | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pioglitazone — Pioglitazone 30 mg o.d. tablet for 12 weeks or placebo o.d. tablet for 12 weeks in random order. After 12 wk treatment there is a 4 wk washout out which is followed by switch of study medication in a cross over fashion and a further 12 wk treatment.

SUMMARY:
The purpose of this study is to test whether pioglitazone is able to prevent the progression of diabetic nephropathy in kidney transplant recipients with diabetes mellitus.

DETAILED DESCRIPTION:
About 30 % of kidney transplant recipients will develop diabetes mellitus. This condition is a risk factor for graft dysfunction, graft loss and increased mortality of patients. Inflammatory reactions within the graft and proteinuria are considered as pathogenetic mechanisms.

Recent studies indicated that pioglitazone might have beneficial effects on the urinary protein excretion of type 2 diabetic patients with diabetic nephropathy and was able to reduce systemic inflammation.

This lead to the hypothesis that pioglitazone could improve proteinuria of kidney transplant patients with diabetes.

Comparison: Effects of pioglitazone vs. placebo on proteinuria and renal function of kidney transplant recipients in a cross over study.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplantation(> 6 months ago) ; stable graft function
* diabetes mellitus type 2
* acceptable glycemia (HbA1c < 8%)
* creatinin clearance (MDRD)>30 ml/min 1,73m²)
* proteinuria > 30 mg/24 hr

Exclusion Criteria:

* type 1 diabetes
* pregnant or breast feeding women
* congestive heart failure (>stage 1 NYHA)
* creeping creatinin
* treatment for rejection within 3 months prior to inclusion
* ALT, AST > 2.5 fold the upper limit of normal
* uncontrolled hypertension
* hypo- or hyperthyroidism

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
proteinuria | 12 weeks

SECONDARY OUTCOMES:
efficacy: filtration fraction, renal nitric oxide bioavailability, insulin resistance, platelet function safety: tolerability, plasma glucose, body weight, edema | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gross, MD, Principal Investigator — Nephrology, Department of Medicine, University hospital Dresden
Locations (1):
- Nephrology, Department of Medicine, university hospital Dresden, Dresden, Germany

REFERENCES:
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882